CLINICAL TRIAL: NCT01405001
Title: Registry of Emergency Airways Arriving at Combat Hospitals (REACH)
Brief Title: Registry of Emergency Airways Arriving at Combat Hospitals
Acronym: REACH
Status: Completed | Type: Observational
Sponsor: William Beaumont Army Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C.2005.055et
Record Dates: First submitted 2011-07-27; First posted 2011-07-28 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Trauma; Wounds and Injuries; Emergencies
Keywords: Emergencies; War; Intubation, Intratracheal
MeSH Terms: conditions — Wounds and Injuries; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This represents the first prospective examination of advanced airway management under combat conditions. The findings will have a tremendous impact on both modern prehospital medical practice and on the treatment of our wounded Soldiers during the Global War on Terrorism.

DETAILED DESCRIPTION:
Stabilizing trauma victims in the out-of-hospital setting often requires the critical intervention of definitive airway management. Prehospital airway management studies in the U.S. have demonstrated variable success with endotracheal intubations by paramedics, ranging from 75-94% in recent well designed studies. Initial prehospital airway efforts showed there was a significant improvement in patient outcome when endotracheal intubation was performed in the field. Yet, a recent review cited 14 studies that demonstrated either no difference or even a higher mortality noted among patients that received prehospital endotracheal intubation by a paramedic. Of note, all of these previous studies were performed in non-combat settings and involved only civilian paramedics.

There currently are no prospective studies in the literature involving prehospital combat advanced airway management. Furthermore, it is not even clear how commonly advanced airway procedures are performed on the modern battlefield. Data from Vietnam shows that 6% of the soldiers killed in action suffered isolated airway injuries. In the current Global War on Terror, an estimated 27% of wounds occur to the head, neck or airway structures. Military databases demonstrate that patients requiring emergency airway management before reaching a combat support hospital constitute 5 to 10% of the total combat casualty population, and that acute airway compromise is a significant cause of preventable traumatic death in modern warfare. During Operation Iraqi Freedom, approximately 10% of the 3600 trauma patients that reached his Combat Support Hospital (CSH) had airway compromise as the primary cause of death. This may represent a conservative estimate given that it is not clear how many patients with airway compromise died on the battlefield and were never transferred to the CSH. In today's world, these findings are important to civilian physicians as well because of the parallels between combat settings and other austere environments such as wilderness medicine, medical support for law enforcement, and managing mass casualty effects of terrorist attacks and weapons of mass destruction.

The purpose of this study was to evaluate advanced airway management performance by prehospital providers during Operation Iraqi Freedom. Our intentions were to provide a preliminary analysis of prehospital airway management within the combat setting, and identify means of improving outcomes associated with prehospital endotracheal intubations. Other points of interest included gaining insight into which providers were at risk for performing incorrect intubations; theorizing how endotracheal intubations could be improved in the combat setting; and comparing the rate of missed intubations to previous studies performed in civilian settings.

This was a prospective, observational study performed under combat conditions during Operation Iraqi Freedom. This study was approved by the U.S. Army Clinical Investigation Regulatory Office. The primary outcome was independently physician verified correct placement of endotracheal tubes by prehospital providers within the combat setting.

ELIGIBILITY:
Inclusion Criteria:

* Casualties presenting to the Combat Support Hospital (CSH) who received advanced prehospital airway on the battlefield.

Exclusion Criteria:

* Casualties who received the initial advanced prehospital airway at the Combat Support Hospital (CSH).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: battlefield casualties who received advanced pre-hospital airway on the battlefield
Enrollment: 292 (Actual)
Dates: Start 2004-12; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Adams, MD, Principal Investigator — William Beaumont Army Medical Center

IPD SHARING:
Plan to Share IPD: Undecided